CLINICAL TRIAL: NCT05830604
Title: Evaluation of the Effect of Muscle Activity on Subjective Tinnitus in Temporomandibular Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Berkan Altay, DDS, DDS, Assist. Prof. Department of Oral and Maxillofacial Surgery, Kutahya Health Sciences University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-09/07
Record Dates: First submitted 2023-03-16; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Tinnitus, Subjective; Temporomandibular Disorder
MeSH Terms: conditions — Tinnitus; Temporomandibular Joint Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TMD Wilkes Stage I-II and Subjective Tinnitus (Active Comparator): Patients with subjective tinnitus and temporomandibular disorder. It was treated with an occlusal splint.
  Interventions: Procedure: Occlusal Splint Treatment- Non Invasive treatment
- TMD Wilkes Stage I-II, Subjective Tinnitus and Bruxism (Active Comparator): Patients with subjective tinnitus and temporomandibular disorder and bruxism. It was treated with an occlusal splint.
  Interventions: Procedure: Occlusal Splint Treatment- Non Invasive treatment

INTERVENTIONS:
Procedure: Occlusal Splint Treatment- Non Invasive treatment — Each patient in the study had temporomandibular disorder. The first-line routine treatment of this disease is an occlusal splint. This treatment was applied to each patient. Surgical intervention was not performed.

SUMMARY:
Treatment of Temporomandibular Joint Disorder can help reduce subjective tinnitus levels. This treatment changes the electrical activity of the patient's chewing muscles. For this reason, the relationship between muscular change and tinnitus levels can be evaluated.

DETAILED DESCRIPTION:
The study will be conducted with patients who routinely apply to Kütahya Health Sciences University Faculty of Dentistry. 70 patients with temporomandibular disease accompanied by tinnitus and bruxism will be included in the study. Demographic data such as age, gender, and systemic disease, drug and trauma history data will be collected.

TMD findings of the patients will be classified according to Wilkes classification. The Wilkes classification is as follows:

1. Stage 1 (early period): No pain or limitation of jaw movements, only reciprocal click during or after chewing. Mild anterior disc displacement in radiological evaluation.
2. Stage 2 (early/intermediate): Mild to moderate pain with reciprocal clicking and periodic locking. Change in disc position.
3. Stage 3 (intermediate): Joint tenderness with frequent pain. Ongoing crash. On the radiological image, changes in disc position and deformation with adhesions.
4. Stage 4 (intermediate/late): Chronic pain that gets worse from time to time and limitation in jaw movements. Change in the shape and position of the disc and the shape of the condyle. Multiple adhesions with hard tissue changes.
5. Stage 5 (late stage): pain that occurs from time to time with crepitation.

Bruxism data (time of onset, whether it is felt during the day/night, fatigue, difficulty in opening the mouth in the morning, stressful period) are questioned and examination findings (disc displacement, masseter hypertrophy on inspection, linea alba, attrition of teeth, fractures in restorations and teeth, muscle and joint pain) , facial asymmetry, mouth opening) will be recorded. The characteristics of tinnitus (objective/subjective, duration, in which ear, increasing and decreasing factors, type) and hearing loss, vertigo will be questioned.

Patients will be divided into two groups. Group I will consist of Wilkes Stage 1-2 patients with temporomandibular intra-articular disorder. Group II will consist of patients with both Wilkes Stage 1-2 temporomandibular intra-articular disorder and bruxism.

In order to measure the muscle strength of the patients before the treatment, EMG containing right-left M. Masseters will be taken in order to easily reach the chewing muscles and to minimize the patient's discomfort. The analog EMG signal will be amplified using a differential amplifier with a high common-mode rejection ratio (bandwidth 5 KHz, peak-to-peak input range 200 μV). The average of the signals is over 500 ms. (Micromed, Italy)

Superficial EMG will be taken following the following protocol:

To reduce skin impedance, the skin will be cleaned before electrode placement and recordings will be made after 5-6 minutes.

Superficial electrodes will be placed on the right and left masseter muscles, with the upper pole of the electrode parallel to the intersection between the tragus-labial commissura and the exocantion-gonion lines. The grounding electrode will be placed in the forehead area.

For all tests, patients will be seated with their head unsupported and asked to maintain a natural upright position.

To avoid any effects of fatigue, a rest period of at least 3 minutes will be allowed between tests. The average EMG potential for each of the muscles will be set to 100%.

To standardize EMG potentials, two 10 mm thick cotton rolls will be placed on each subject's mandibular first and second molars, and maximum voluntary clamping of 5 seconds will be recorded. For 5 seconds, the patient will be encouraged to maintain the same level of contraction. EMG data analysis for all tests, the best 3-s period (the one with the most stable signal) will be automatically selected by the software and used for all subsequent analysis.

Electromyographic activity will then be recorded with a maximum voluntary squeeze at the intercuspal position; The patient will be invited to squeeze as hard as possible and maintain the same level of contraction for 5 seconds. Electromyographic activity will also be taken again while the patient is at rest.

For each subject, the EMG potentials of the analyzed muscles recorded during the maximum voluntary clamping tests will be expressed as a percentage of the average potential recorded during the standardization test (maximum voluntary clamping on cotton rolls).

(μV/μV×100). To assess muscle symmetry, the EMG waves of the masseter muscles will then be compared by calculating a percent overlap coefficient (POC, %). POC is an index of the symmetrical distribution of muscle activity determined by occlusion. The index ranges from 0% to 100%: a POC of 100% will be achieved when two paired muscles contract with perfect symmetry.

Tinnitus and bruxism will be evaluated by the patient with the VAS score. Tinnitus level will additionally be measured with the Tinnitus Handicap Inventory. Then, an occlusal splint will be prepared for the patients. It will be recommended to use them for 24 weeks. Postoperative EMG, Tinnitus Handicap Inventory and VAS scores will be re-evaluated after the use of the occlusal splint.

The obtained data beam when; Age, gender, disease findings, preoperative and postoperative Tinnitus Handicap Inventory and VAS scores, masseter and temporal muscle strength in EMG will be compared and evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Patients with chronic subjective tinnitus
* Patients with Wilkes Stage 1-2

Exclusion Criteria:

* Patients with Wilkes Stage 3-4-5
* Patients with tinnitus due to audiological, neurological, metabolic or pathological reasons
* Patients with objective tinnutus
* Patients with normal tinnitus
* Mentally retarded patients
* Hearing loss, use of ototoxic drugs
* Those with ear diseases such as acute ostitis media, perforated tympanic membrane
* Those with Meniere's disease
* Patients with middle ear pathology
* Those with intracranial pathology
* Those with traumatic cervical spine injury
* Patients with severe depression diagnosed by a psychologist
* Patients who have received TMB treatment in the last two months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
Masseters Activity | 6th months
  To evaluate the symmetry and electrical activity of masseters by surface EMG

CONTACTS AND LOCATIONS:
Overall Officials: Elif Çoban, DDS, Principal Investigator — https://avesis.ksbu.edu.tr/elif.coban/iletisim; Mehmet Ç. Ulucan, DDS, Principal Investigator — https://avesis.ksbu.edu.tr/mehmetcagatay.ulucan; Selver S. Başak, DDS, Principal Investigator — https://avesis.ksbu.edu.tr/selversuna.basak; Berceste Güler, DDS, Principal Investigator — https://avesis.ksbu.edu.tr/berceste.guler; Merve Akdeniz Leblebiciler, MD, Principal Investigator — https://avesis.ksbu.edu.tr/merve.akdenizleblebicier; Vural Kavuncu, MD, Principal Investigator — https://avesis.ksbu.edu.tr/vural.kavuncu
Locations (1):
- Kütahya Health Science University, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-20): https://cdn.clinicaltrials.gov/large-docs/04/NCT05830604/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-20): https://cdn.clinicaltrials.gov/large-docs/04/NCT05830604/ICF_001.pdf